CLINICAL TRIAL: NCT07033377
Title: Cross-Cultural Adaptation and Psychometric Validation of the Persian Version of the Cognitive Behavioral Questionnaire in Nonspecific Chronic Low Back Pain
Brief Title: Psychometric Validation of Persian CBQ-NSCLBP
Status: Not yet recruiting | Type: Observational
Sponsor: Kourosh Najafi (Other)
Responsible Party: Sponsor-Investigator, Kourosh Najafi, MSc Student, Department of Physiotherapy and Rehabilitation, Medipol University
Organization: Medipol University (Other)
Other Study IDs: MEDI-CBQNSCLBP-Pe
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Nonspecific Chronic Low Back Pain
Keywords: chronic low back pain; CBQ-NSCLBP; Persian version; cross-cultural adaptation; psychometric validation; CLBP; cognitive behavioral questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-administered paper-based questionnaires — Participants will complete the Persian version of the CBQ-NSCLBP and other self-report measures as part of a psychometric validation study. No clinical or therapeutic intervention is involved.

SUMMARY:
This study aims to translate, culturally adapt, and psychometrically validate the Persian version of the Cognitive Behavioral Questionnaire in Nonspecific Chronic Low Back Pain (CBQ-NSCLBP). The process will follow standard cross-cultural adaptation guidelines, including forward-backward translation, expert review, and pilot testing. The psychometric properties, including internal consistency, test-retest reliability, and construct validity, will be evaluated in a sample of Persian-speaking adults with nonspecific chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a common and persistent musculoskeletal condition that affects a large portion of the population and can lead to long-term disability. It is typically defined as pain in the lower back that lasts for more than 12 weeks and often impacts daily function and quality of life.

In addition to physical symptoms, people with CLBP frequently experience cognitive and behavioral challenges, such as fear-avoidance beliefs, catastrophizing, and difficulty concentrating. These factors can contribute to ongoing disability and interfere with the rehabilitation process.

The Cognitive Behavioral Questionnaire for Nonspecific Chronic Low Back Pain (CBQ-NSCLBP) was developed to assess these cognitive-behavioral aspects in people with nonspecific CLBP. However, it has only been validated in one population and has not yet been adapted for Persian-speaking individuals.

This study aims to translate and culturally adapt the CBQ-NSCLBP into Persian and evaluate its psychometric properties in individuals with nonspecific chronic low back pain

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 65 years old.
* Experiencing nonspecific low back pain for at least 6 months.
* Have a physician-confirmed diagnosis.
* Be able to read and understand Persian.
* Be willing to participate and provide written informed consent.

Exclusion Criteria:

* Specific causes of low back pain (e.g., spinal infection, tumor, fracture, inflammatory disease, radiculopathy, or other neurological disorders).
* Severe psychiatric disorders or cognitive impairments interfering with questionnaire comprehension.
* History of surgery for low back pain.
* Abnormal bowel or bladder function.
* Pregnant at the time of participation.
* Not fluent in Persian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years diagnosed with nonspecific chronic low back pain by a physician, who are fluent in Persian and able to complete questionnaires independently. Participants will be recruited from physiotherapy clinics and outpatient rehabilitation centers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CBQ-NSCLBP | Baseline and within 6 to 10 days after enrollment
  Evaluation of the internal consistency, test-retest reliability, and construct validity of the Persian version of the Cognitive Behavioral Questionnaire in Nonspecific Chronic Low Back Pain (CBQ-NSCLBP).

IPD SHARING:
Plan to Share IPD: No